CLINICAL TRIAL: NCT05138198
Title: Lifestyle Intervention to Reduce Body Weight and Systemic Inflammation Among World Trade Center Responders With PTSD: Pilot Randomized Controlled Trial
Brief Title: Lifestyle Intervention to Reduce Body Weight and Systemic Inflammation Among World Trade Center Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Chrisa Arcan, PhD, MHS, MBA, RD, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: U01OH012057 (NIH)
Record Dates: First submitted 2021-08-07; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Post-Traumatic Stress Disorder; Overweight and Obesity; Metabolic Syndrome; Inflammation
Keywords: Post-Traumatic Stress Disorder; Overweight and Obesity; Inflammation; Mediterranean Diet; Physical Activity; World Trade Center Responders; Metabolic Syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Overweight; Obesity; Metabolic Syndrome; Inflammation; Motor Activity | interventions — Diet, Mediterranean; Exercise; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet & Physical Activity (Experimental): Nutrition with a Physical Activity component. 10-week intervention implementing the Mediterranean Diet.
  Interventions: Behavioral: Mediterranean Diet & Physical Activity
- Usual Care (Active Comparator): Usual care involves one-on-one monthly nutrition counseling
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Mediterranean Diet & Physical Activity — At the beginning of each week (1-10), members were sent a text message introducing the week and providing the link to the week's website. This website includes downloadable material for this group with recipes and other important nutrition information, as well as the weekly topic information and informative video. After receiving the link to the website, members received a Qualtrics survey with a teach-back question related to the video and a goal-setting question related to the topics of the week. At the end of each week, members received another Qualtrics survey with a question regarding the goal of the past week.
  * Visit 1: discuss Mediterranean diet score results from baseline and ways to improve
  * Visit 2: discuss anti-inflammatory diet scorecard and ways to improve
  * Discuss optimal dietary pattern (Med Diet pyramid handout)
  * Personal dietary and exercise goals, reviewed baseline intake form, social support, self-efficacy, challenges, or barriers to achieving goals
  Other Names: Nutrition Intervention
  Arms: Mediterranean Diet & Physical Activity
Behavioral: Usual Care — As part of usual care, members attended one-on-one monthly counseling sessions with the assigned dietitian and reviewed their current eating habits and physical activity, as well as other environmental factors that may be affecting their weight such as work, home environment, sleeping issues, and medications. After reviewing current practices, the RD provided medical nutrition therapy (MNT), a specific application of the Nutrition Care Process in clinical settings that focuses on the management of diseases (e.g. diabetes, heart disease, etc.). Specific dietary recommendations are based on the Bull's Eye Food Guide, used by Stony Brook University Hospital for outpatient nutrition counseling. Individuals in the standard care received more individualized calorie recommendations (usual care) than the Mediterranean diet group.
  Other Names: Control
  Arms: Usual Care

SUMMARY:
The goal of this randomized control trial (RCT) is to test the feasibility and acceptability of a lifestyle intervention with a focus on implementing a high dose Mediterranean Diet protocol with physical activity to reduce systemic inflammation and body weight among WTC first responders having overweight/obesity and PTSD. The findings of this study will demonstrate the suitability of the proposed approach to reduce comorbidities among similar populations exposed to traumatic events; the findings will also inform the World Trade Center Health Program's extensive research and clinical efforts with the potential to provide a preventive care model to reduce systemic inflammation and related chronic disease among WTC responders with PTSD.

DETAILED DESCRIPTION:
The proposed study will assess the feasibility and acceptability of a lifestyle intervention, including a Mediterranean Diet (MedDiet) with a physical activity (PA) component. The study is a pilot randomized control trial (RCT) among WTC responders with PTSD who have overweight and obesity. The 10-week intervention has two-arms, the intervention (MedDiet) with tips to increase PA (n=30) and control (care as usual n=30).

The high dose and high fidelity intervention combines several previously tested intervention modalities, including individual nutrition counseling, group cooking sessions, and communication and education through smartphones, including motivational texts & reminders, videos, teach-back surveys, and goal setting. While the main goal of the intervention is to assess the feasibility and acceptability of the intervention, the study will also assess changes in the overall dietary intake, the MedDiet score, and PA of the intervention group and between the two groups from baseline, post-intervention, and 3-month follow-up. The hypothesis is that the intervention group will experience a significant increase in the MedDiet score and PA activity from baseline to post-intervention; compared to the control group, the intervention group will achieve a significantly higher MedDiet score and will engage in more PA after the intervention.

Changes in body weight, inflammatory biomarkers, and prevalence of metabolic syndrome (MetS) in the intervention group and between the two groups from baseline to post-intervention will be explored; whether changes in inflammatory biomarkers, are moderated by changes in MetS, body weight, or MedDiet score will also be explored. The hypothesis is that the intervention group will experience a significant decrease in inflammatory biomarkers and prevalence in MetS from baseline to post-intervention; compared to the control group, the intervention group will achieve a significantly higher decrease in these measures; the decline in inflammatory biomarkers will be moderated by a reduction in the prevalence of MetS and/or increase in MedDiet score.

ELIGIBILITY:
Inclusion Criteria:

* BMI range: 27-40
* PCL score: ≥40
* MOCA score: ≥22
* have a smartphone
* able to follow a diet intervention
* no physical disabilities which prevent exercising

Exclusion Criteria:

* active cancer or history of GI-related cancer in the last 3 years
* autoimmune disease
* history of surgical weight loss

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Mediterranean diet score | 9 months
  Participant's Mediterranean diet score is measured with a 14-item Mediterranean diet scale; possible score range 0-14.
  The Mediterranean Diet questionnaire will be given at each participant visit with the dietitians and at baseline, post, and at 3-month follow up

SECONDARY OUTCOMES:
Physical activity | 9 months
  Daily step count is measured with Fitbit that was worn over seven days. Physical activity are measured at baseline, post-intervention, and 3-month follow up.
Body mass index (BMI) | 9 months
  Body mass index (weight/height square) will be objectively measured at baseline, post intervention and at 3-month follow up.
  Body mass index: weight in kilograms/square of height in meters
Waist Circumference | 9 months
  Waist circumference is measured at baseline, post-intervention, and 3-month follow up.
  Waist circumference cut off (Women>88cm; Men>102 cm)
Total cholesterol | 9 months
  Total cholesterol is measured at baseline, post-intervention, and at 3-months follow-up; reference range: 125 to 200mg/dL
oxidized LDL | 9 months
  Serum oxLDL is measured at baseline, post-intervention, and at 3-months follow-up; reference range: 10-170 ng/mL
HDL cholesterol | 9 months
  Serum HDL cholesterol was measured at baseline, post-intervention, and at 3-months follow-up;
  At risk Men: Less than 40 mg/dL (1.0 mmol/L) Women: Less than 50 mg/dL (1.0 mmol/L)
Omega 3 fatty acid | 9 months
  Serum or plasma Free (Nonester) Fatty Acids Measured at baseline, post-intervention, and at 3-months follow-up. reference range:
  Optimal >3.2 % Moderate 2.2-3.2 % High <2.2 %
Omega 6 to omega 3 ratio | 9 months
  Omega 6 is measured at baseline, post-intervention, and at 3-months follow-up;
  Omega 6/omega 3 ratio:
  Reference range: 5.7-21.3 (the lower the better)
HA1c | 9 months
  Serum Hemoglobin A1C (hA1C) is measured at baseline, post-intervention, and 3-month follow up.
  hA1C: Normal: <5.7%
Cytokines | 6 months
  The following cytokines will be measured:
  FNɣ, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-22 and TNFα, high-sensitivity C-reactive protein (hs-CRP) at >3mg/L.
  The cytokines will be measured at two time points at baseline and post-intervention.
Psychosocial questionnaire | 9 months
  A total of 40 questions will be used to assess sedentary behaviors, home food availability, social support, self-efficacy, perceived barriers to adhering to lifestyle behaviors reflecting the behavioral strategies that will be addressed in the proposed intervention. The survey will be completed online at baseline, post-intervention and at 3-month follow up.
PCL score | 9 months
  Post Traumatic Stress Disorder symptoms will be tested with a PCL score. PCL is a 20-item self-report measure of current (past month) PTSD symptoms based on the DSM-V criteria. PCL will be measured at baseline, post intervention and at 3-month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- World Trade Center Health Program Clinic, Commack, New York, United States